CLINICAL TRIAL: NCT00807404
Title: Forward Image Guided Ductoscopy for Early Cancer Screening
Brief Title: Optical Coherence Tomography in Tissue Samples From Women Undergoing Mastectomy for the Treatment or Prevention of Breast Ductal Intraepithelial Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000628769; P30CA033572 (NIH); CHNMC-06008
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Precancerous Condition
Keywords: ductal intraepithelial neoplasia
MeSH Terms: conditions — Precancerous Conditions | interventions — Tomography, Optical Coherence

INTERVENTIONS:
Procedure: histopathologic examination
Procedure: optical coherence tomography

SUMMARY:
RATIONALE: New diagnostic procedures, such as optical coherence tomography, may be effective in finding tumor cells.

PURPOSE: This clinical trial is studying optical coherence tomography in tissue samples from women undergoing mastectomy for the treatment or prevention of breast ductal intraepithelial neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To design and construct a portable forward imaging optical coherence tomography (OCT) needle probe.
* To compare OCT imaging of ex-vivo breast tumor tissue sections with histology to form the basis of an image library for in-vivo work.
* To initiate development of an OCT needle probe that is capable of acquiring core biopsy samples.

OUTLINE: Breast tissue samples are obtained during mastectomy and analyzed ex-vivo by optical coherence tomography (OCT) and by histopathological examination. Once routine pathological evaluation and tissue sampling are completed, OCT imaging is performed using a portable forward imaging needle probe that is inserted through the ducts of the tissue sample. OCT images of the surface of the closest margin to the tumor (if present) as well as images of the duct(s) in the nipple areola complex (after dilation) are obtained. Images of a cross section of the tumor (after the sample has been sliced by the pathologist) are also obtained. The OCT images are then correlated with tissue histology. The images are used to create a correlation histology-OCT atlas for the evaluation of subsequent images and for future reference.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing mastectomy at the City of Hope Breast Center for the treatment or prevention of breast ductal intraepithelial neoplasia

PATIENT CHARACTERISTICS:

* Fertile and/or pregnant patients allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Design of a portable forward imaging optical coherence tomography (OCT) needle probe
Comparison of OCT imaging of ex-vivo breast tumor tissue sections with histology
Development of an OCT needle probe that is capable of acquiring core biopsy samples

CONTACTS AND LOCATIONS:
Overall Officials: I. B. Paz, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States